## **Study Protocol – Cover Page**

Official Title of the Study: The Effect of Kinesiologic Taping on Trunk Control and

Balance in Children with Cerebral Palsy

**NCT Number:** NCT0XXXXXXX

**Document Type:** Study Protocol

**Document Date: August 1, 2025** 

Principal Investigator: Dr. Özden Baskan

Istanbul Rumeli University/ The Department of Physical Therapy and Rehabilitation

Address: Istanbul Rumeli University Kadıköy Campus

Bostancı, Tünel Girişi Street No:10 34744 Kadıköy / Istanbul, Turkey ozdenbaskan@gmail.com

Sponsor / Collaborator: Istanbul Rumeli University

This study did not receive any external funding and was conducted within Istanbul Rumeli University.

## The Effect of Kinesiologic Taping on Trunk Control and Balance in Children with Cerebral Palsy

**Background:** This pre-post, single-group clinical study evaluates the effects of kinesiology taping on motor function, balance, spasticity, trunk control and joint range of motion in children with hemiplegic or diplegic cerebral palsy over a period of four weeks.

**Objective:** This study aims to investigate the effect of kinesiologic taping (KT) on body control and balance in children with spastic cerebral palsy.

Methods: Children with spastic cerebral palsy (aged 2 to 18 years) who have attended regular physiotherapy sessions for at least six months and have a Gross Motor Function Classification System (GMFCS) level of 1, 2, or 3 will be included. The study includes pre- and post-intervention assessments using Range of Motion (ROM), Gross Motor Function Classification System (GMFCS), Functional Independence Measure for children (WeeFIM), Paediatric Berg Balance Scale (PBS), Sitting Assessment Scale (SAS), manual muscle testing of the trunk (MMT), and spasticity assessment using the Modified Ashworth Scale (MAS). Participants will be evaluated at the beginning and end of the fourth week. Taping will be performed four times in total, once a week.

**Ethical Approach:** All procedures conform to the ethical standards of the Helsinki Declaration and were approved by the Istanbul Rumeli University Human Subjects Protection Review Board (Approval No: 2024/08 item:17).

**The Statistical analysis:** Analysis will be performed using [e.g., paired t-tests or appropriate non-parametric tests] to evaluate within-group changes from pre- to post-intervention.